CLINICAL TRIAL: NCT04379102
Title: The Role Of Local Anesthetics Effects During Intrauterine Device Application
Brief Title: The Role Of Local Anesthetics in the Management of Adverse Effects Associated With Intrauterine Device Application
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: ntria
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: IUD; Contraception; Pain
MeSH Terms: conditions — Pain | interventions — Therapeutics; Anesthetics, Local; thymus-leukemia antigens

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IUD patients: 80 patients who matched the inclusion criteria and received IUDs
  Interventions: Other: with NT/TLA (NT or also referred to as therapy with local anesthetics (TLA) )

INTERVENTIONS:
Other: with NT/TLA (NT or also referred to as therapy with local anesthetics (TLA) ) — Patients who visited our family planning clinic and opted for IUD application for contraception purposes were also offered NT/TLA treatments simultaneously. 40 patients who matched the inclusion criteria and received IUDs and NT/TLA treatments were included in the study group and 41 patients who only received IUDs were included in the control group. All patients received copper IUDs and none of them were on additional hormonal treatment. Before the insertion of IUD, women in the therapy group received NT treatment with 6ml of 1% procaine injected transvaginal into the cervix at 5 and 7 o'clock localizations.
  Other Names: without NT/TLA (NT or also referred to as therapy with local anesthetics (TLA) )

SUMMARY:
Patients who visited our family planning clinic and opted for IUD application for contraception purposes were also offered NT/TLA treatments simultaneously. 40 patients who matched the inclusion criteria and received IUDs and NT/TLA treatments were included in the study group and 41 patients who only received IUDs were included in the control group. All patients received copper IUDs and none of them were on additional hormonal treatment. Before the insertion of IUD, women in the therapy group received NT treatment with 6ml of 1% procaine injected transvaginal into the cervix at 5 and 7 o'clock localizations. Following IUD insertion, another 6ml of 1% procaine was injected into the Frankenhauser ganglia bilaterally. A final dose of 8ml of 1% procaine was injected into the abdominal trigger points and intracutaneously into the L4-S4 dermatomes as quaddles.

ELIGIBILITY:
Inclusion Criteria:

* not pregnant women
* healty women age between 18- 45 years old

Exclusion Criteria:

* chronic diseases which could cause chronic pelvic pain such as endometriosis
* which makes them prone to infections such as diabetes mellitus
* complication had arised during the IUD insertion, such as uterine perforation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women with underlying chronic diseases which could cause chronic pelvic pain such as endometriosis and which makes them prone to infections such as diabetes mellitus were excluded from the study. Furthermore, women by whom a complication had arised during the IUD insertion, such as uterine perforation, were also excluded from the study.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
The VAS scores of patients after the application of IUDs | 1 month
  The VAS scores of patients in both groups reported one month after the application of IUDs (Patients mark their pain intensity from 1 to 10 in vas scoring. In scoring, 1 point is the lowest score and shows that the patient has low pain, 10 is the highest score and shows severe pain.)

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes